CLINICAL TRIAL: NCT04578457
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - 2020_09
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2020_09
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hearing Aid without NR(0) enabled (Active Comparator): Hearing Aid without Noise Reduction (NR 0) enabled serves as reference condition.
  Interventions: Device: Hearing Aid without NR enabled
- Hearing Aid with NR (1) (Experimental): Hearing Aid with Noise Reduction I (NR) enabled.
  Interventions: Device: Hearing Aid with NR(1)
- Hearing Aid with NR(2) (Experimental): Hearing Aid with Noise Reduction II (NR) enabled.
  Interventions: Device: Hearing Aid with NR(2)
- Hearing Aid with NR(3) (Experimental): Hearing Aid with Noise Reduction III (NR) enabled.
  Interventions: Device: Hearing Aid with NR(3)

INTERVENTIONS:
Device: Hearing Aid without NR enabled — Each participant will be fitted with noise reduction disabled. Disabled means that no sound processing algorithm that removes noise from the speech signal is active.
  Arms: Hearing Aid without NR(0) enabled
Device: Hearing Aid with NR(1) — Each participant will be fitted with the noise reduction program on the same hearing aid. The principle of the noise reduction algorithm is to remove noise from a speech signal with the aim of improving the speech intelligibility and comfort.
  Arms: Hearing Aid with NR (1)
Device: Hearing Aid with NR(2) — Each participant will be fitted with a second noise reduction program on the same hearing aid. The parameterization of this NR algorithm differs from that in NR(1).
  Arms: Hearing Aid with NR(2)
Device: Hearing Aid with NR(3) — Each participant will be fitted with a third noise reduction program on the same hearing aid. The parameterization of this NR algorithm differs from that in NR(1) and NR(2).
  Arms: Hearing Aid with NR(3)

SUMMARY:
Participants will perform two different listening tasks: (1) listening to, and repeating back, sentence lists presented in noise, and (2) Subjective rating of effort & performance following each condition. During this study, continuous, non-invasive physiological measurements (skin conductance, changes in pupil dilation) will be recorded from participants. Using this paradigm we will be assessing the effect of different hearing aid processing algorithms on listening effort. The study takes the form of a one factor (algorithm), within-subjects design.

Each participant performs the Speech perception task with each algorithm (reference, noise reduction I, noise reduction II, noise reduction III), at two individualized signal-to-noise ratios (SRT90 and SRT50). Additionally subjective performance ratings in real-life will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature
* Minimum 1 year hearing aid experience
* Moderate-Severe (N3-N5) hearing loss or Normal Hearing

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Condition: This was a crossover "within subject design" study in which all participants undertook all study conditions.
  These conditions consisted of different hearing aid settings, and were interleaved within study appointments.
  Accordingly, the different conditions are reported here as study 'Periods' to avoid participants being included multiple times in the overall protocol count.
  This means there will be a discrepancy whereby the number starting a period will be greater than the number completing the previous 'period'. Of course this is simply due to the fact that the study 'periods' as reported are not chronological.
Period: Hearing Aid Without NR Enabled (0)
Arm/Group | Randomized Condition
Started | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Hearing Aid With NR (1)
Arm/Group | Randomized Condition
Started (The discrepancy between the number of participants starting this period and finishing the previous period is simply due to the fact that the study 'periods' as reported are not chronological. See 'Arm/Group Description' for details.) | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Hearing Aid With NR (2)
Arm/Group | Randomized Condition
Started (The discrepancy between the number of participants starting this period and finishing the previous period is simply due to the fact that the study 'periods' as reported are not chronological. See 'Arm/Group Description' for details.) | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Hearing Aid With NR (4)
Arm/Group | Randomized Condition
Started (The discrepancy between the number of participants starting this period and finishing the previous period is simply due to the fact that the study 'periods' as reported are not chronological. See 'Arm/Group Description' for details.) | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Cohort: This study was a crossover design, therefore there was only a single study group.
  This group undertook measures under each of the study conditions.
Arm/Group | Study Cohort
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.95 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 19

OUTCOME MEASURES:

1. Primary Outcome: Differences in Event-related-skin-conductance
Description: Skin conductance will be recorded from participants during the performance of the auditory task. Analyses will be carried out on the skin conductance response recorded during a time window following each auditory stimulus. It is planned to analyze event-related skin conductance response amplitudes & latencies (micro-Siemens & milliseconds).
Time Frame: 6 weeks
Population: The data from some participants had to be excluded from the analysis. Due to the noisy nature of physiological data, in some cases we were unable to collect enough valid, artefact-free data to analyse. Where this was the case, we discounted the participant from analyses. As we only contrasted NR(0) vs NR(1) and NR(2) vs NR(3) (and collected respective data at different study appointments), there is a slight discrepancy in the number of participants analysed for these study arms.
Measure: Mean (95% Confidence Interval); unit: micro Siemens
Arm/Group | Hearing Aid Without NR(0) Enabled | Hearing Aid With NR (1) | Hearing Aid With NR(2) | Hearing Aid With NR(3)
Number analyzed (Participants) | 15 | 15 | 16 | 16
micro Siemens | 0.221 [0.176 to 0.267] | 0.189 [0.150 to 0.227] | 0.147 [0.099 to 0.195] | 0.126 [0.099 to 0.153]

2. Primary Outcome: Differences in Event-related-pupil-dilation (ERPDs)
Description: Pupil dilations will be recorded from the participant during the performance of the auditory tasks.
  Analyses will be carried out relative to the pre-trial baseline (measured one second prior to the onset of the stimulus), in order to account for differences in baseline physiological activity.
  It is planned to analyze event-related-pupil-dilations. We use the unit: pixels. The size of a pixel in 1mm^2 is relative to the distance between the eye and the camera. Even though participants heads were placed on a chin rest that was always the same distance from the camera, the distance between the individual eye and the camera can still be different due to differences in participants' anatomies.
  Thus, pupil dilation are often reported relative to an individuals' baseline, for example as percent change relative to the baseline.
  Therefore, we use the unit: pixels, as the use of mm^2 may be inaccurate.
Time Frame: 6 weeks
Population: The data from some participants had to be excluded from the analysis. Due to the noisy nature of physiological data, in some cases we were unable to collect enough valid, artefact-free data to analyse. Where this was the case, we discounted the participant from analyses.
Measure: Mean (95% Confidence Interval); unit: pixels
Arm/Group | Hearing Aid Without NR(0) Enabled | Hearing Aid With NR (1) | Hearing Aid With NR(2) | Hearing Aid With NR(3)
Number analyzed (Participants) | 11 | 11 | 11 | 11
pixels | 217.713 [154.747 to 280.689] | 217.301 [164.876 to 269.726] | 158.732 [113.199 to 204.265] | 186.526 [119.151 to 253.900]

3. Secondary Outcome: Oldenburg Sentence Test
Description: Words recalled correctly: words repeated back by participants are logged and the percentage of words recalled correctly calculated.
Time Frame: 6 weeks
Population: By the time this outcome measure was performed, 1 of the original participants had withdrawn from the study.
  Therefore, data for 18 participants was analysed.
Measure: Mean (Standard Deviation); unit: Percentage of correct words
Arm/Group | Hearing Aid Without NR(0) Enabled | Hearing Aid With NR (1) | Hearing Aid With NR(2) | Hearing Aid With NR(3)
Number analyzed (Participants) | 18 | 18 | 18 | 18
Percentage of correct words | 92.778 (3.296) | 88.611 (6.709) | 96.157 (2.271) | 94.398 (4.607)

4. Secondary Outcome: Sound Quality Ratings
Description: The sound quality ratings will be assessed with the aid of a Multi-Stimulus Test.
  The data, serving as secondary outcome measure, are collected in the laboratory.
  The scale ranges from 0 "very bad" to 6 "very good" in increments of 1. Individual sound quality rating from participants are averaged over 3 different acoustic scenes for each hearing aid program.
Time Frame: 6 weeks
Population: By the time this outcome measure was performed, 2 of the original participants had withdrawn from the study.
  Therefore, data for 17 participants was analysed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hearing Aid Without NR(0) Enabled | Hearing Aid With NR (1) | Hearing Aid With NR(2) | Hearing Aid With NR(3)
Number analyzed (Participants) | 17 | 17 | 17 | 17
score on a scale | 3.275 (0.263) | 3.230 (0.107) | 3.054 (0.208) | 3.157 (0.136)

5. Secondary Outcome: Spectro-temporal-modulation Detection Thresholds (STM)
Description: Stimuli which contain simultaneous frequency and amplitude modulations of a wide-band noise carrier are presented to the participants.
  The depth of the modulations is systematically varied and the individual modulation detection thresholds are recorded as a broadband decibel (dB) value.
  For each participant 4 measures were made and averaged to give a mean STM threshold.
Time Frame: 6 weeks
Population: By the time this outcome measure was performed, 2 of the original participants had withdrawn from the study.
  Therefore, 17 participants had measurements for this outcome measure made. For 5 participants it was not possible to measure an STM threshold reliably at all test occasions.
  Where this was the case, these participants were excluded from analyses.
Measure: Mean (Standard Error); unit: decibel
Groups:
- Study Cohort: This was a measure of underlying auditory function. Accordingly it was made without the use of hearing aids (i.e. under a single unaided condition).
  Therefore, the results are reported as a single group.
Arm/Group | Study Cohort
Number analyzed (Participants) | 12
decibel | -8.181 (0.617)

6. Other Pre Specified Outcome: Non-verbal Trail Making Test A & B
Description: The Trail Making Test (TMT) is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible according to a given order. In version A the order is given by increasing digit number (i.e. 1-25) while in version B the order is given by alternating digits and letters (i.e. 1-A-2-B-3-C…). The data, serving as an outcome measure, are time-to-complete the set in seconds.
Time Frame: 2 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Digit-Span Test Forward (FW) & Backward (BW)
Description: The digit-span task is used to measure working memory's number storage capacity. Participants will see a sequence of numerical digits and are tasked to recall the sequence correctly, with increasingly longer sequences being tested in each trial. The participant's span is the longest number of sequential digits that can accurately be remembered, which means that the participant recalls two sequences out of a maximum of three sequences correct. Digit-span tasks can be given forwards or backwards, meaning that once the sequence is presented, the participant is asked to either recall the sentence in normal or reverse order.
Time Frame: 2 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Go/No-go Task
Description: The Go/No-go task measures inhibitory control. Participants are asked to respond to a Go stimulus as fast as possible but not respond to a No-go stimulus. Go stimuli are presented at a rate much higher than the No-go stimuli to elicit prepotent motor activity. The outcome measure of this task is the number of commission errors (i.e. responding to a No-go stimuli) a participant commits as a measure of their ability to stop prepotent motor activity.
Time Frame: 6 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Blood Volume Pulse
Description: Blood volume pulse will be recorded from participants during the performance of the auditory task (non-invasively with a photoplethysmographic (PPG) sensor). Analyses will be carried out on the data recorded during a time window following each auditory stimulus (relative to baseline activity). It is planned to analyze event-related changes in pulse rate and amplitude (beats per minute).
Time Frame: 6 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Respiration Data
Description: Respiration rates will be recorded from participants during the auditory task using a belt placed under the ribcage. This data will only be used to control for changes in breathing patterns which may influence skin conductance measurements.
Time Frame: 6 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Skin Temperature Data
Description: Skin temperature will be recorded from participants during the auditory task using a small thermometer attached to the outside of the little finger (non-dominant hand). This data will only be used to control for changes in temperature which may influence skin conductance measurements.
Time Frame: 6 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Acoustic Reflex Thresholds
Description: Tympanometry will be used to assess the mobility of the eardrum, prior to recording Acoustic Reflex Thresholds (ARTs). Compliance [ml], Middle Ear Pressure [daPa] and ear canal volume [ml] will be recorded and checked that they fall within normal limits. Where this is the case, ARTs will be measured using 0.5, 1 & 2 kHz stimulus tones ipsi- and contralaterally for each ear. The resulting outcome measure will be the threshold [dB] required at each frequency and ear arrangement for a stapedial reflex to be present.
Time Frame: 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Description: This study was a crossover design, therefore there was only a single study group.
  This group undertook measures under each of the study conditions. These conditions were undertaken in an interleaved fashion during the same study appointment.
  As such it is not possible to attribute the adverse event reported to any single condition.
  We therefore report the adverse events here as a function of the entire study population.
Groups:
- Study Cohort: This study was a crossover design, therefore there was only a single study group.
  This group undertook measures under each of the study conditions. These conditions were undertaken in an interleaved fashion during the same study appointment.
  As such it is not possible to attribute the adverse event reported to any single condition.
  We therefore report the adverse events here as a function of the entire study population.
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Cohort (N=19)
Positive test for COVID-19 (General disorders) | 1 — A single participant tested positive for COVID-19 between measurement appointments. This was deemed not to be related to the investigational device or experimental protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04578457/Prot_SAP_000.pdf